CLINICAL TRIAL: NCT02260492
Title: Clinical Endpoint Study of Salmeterol Xinafoate/Fluticasone Propionate Combination for Comparison of a Test and Reference Product in Patients With Asthma
Brief Title: Clinical Efficacy Study of Salmeterol Xinafoate/Fluticasone Propionate in Asthma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oriel Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: OTT329/305
Record Dates: First submitted 2014-10-06; First posted 2014-10-09 (Estimated); Results first posted 2017-06-15 (Actual); Last update posted 2017-06-15 (Actual); Status verified 2017-03

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Salmeterol Xinafoate; Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- OT329 Solis (Experimental): OT329 Solis (twice daily inhalation throughout the study)
  Interventions: Drug: OT329 (combination of fluticasone propionate and salmeterol xinafoate)
- Advair Diskus (Active Comparator): Advair Diskus (twice daily inhalation throughout the study)
  Interventions: Drug: Advair Diskus (combination of fluticasone propionate and salmeterol xinafoate)
- Placebo (Placebo Comparator): Placebo (twice daily inhalation throughout the study)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OT329 (combination of fluticasone propionate and salmeterol xinafoate) — Fluticasone propionate (100 mcg) and salmeterol xinafoate (50 mcg) administered by Solis dry powder inhaler
  Arms: OT329 Solis
Drug: Advair Diskus (combination of fluticasone propionate and salmeterol xinafoate) — Fluticasone propionate (100 mcg) and salmeterol xinafoate (50 mcg) administered by Diskus dry powder inhaler
  Arms: Advair Diskus
Drug: Placebo — Placebo (lactose) administered via the Solis dry powder inhaler
  Arms: Placebo

SUMMARY:
This is a study to establish the equivalence of OT329 Solis and Advair Diskus when administered by inhalation in patients with asthma.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥ 18 years old of non-child bearing potential or of child bearing potential committing to consistent and correct use of an acceptable method of birth control
2. Subjects with a reliable clinical history of asthma documented at least 12 weeks prior to screening
3. Subjects with a pre-bronchodilator FEV1 of > 40% and <85% of the predicted value during the screening visit and on the first day of treatment
4. Subjects who are currently non-smoking and have not used tobacco products (i.e., cigarettes, cigars, pipe tobacco) within the past year, and had < 10 pack-years of historical use
5. Subjects with > 15% reversibility of FEV1 within 30 minutes following 360 mcg of albuterol inhalation (pMDI). Note: This test may be repeated on a different day if the patient fails the first attempt; and if the patient achieves at least 10% reversibility and the Investigator thinks that a second attempt is appropriate
6. Subjects who are able to discontinue their asthma medications (inhaled corticosteroids and long-acting beta agonists) during the run-in period and for the remainder of the study
7. Subjects who are able to replace current short-acting beta agonists (SABAs) with salbutamol/albuterol inhaler for use as needed for the duration of the study (subjects should be able to withhold all inhaled SABAs for at least 6 hours prior to lung function assessments on study visits)
8. Subjects who are able to continue the following medications without a significant adjustment of dosage, formulation, or dosing interval for the duration of the study, and judged able by the investigator to withhold them for the specified minimum time intervals prior to each clinic visit: short-acting forms of theophylline for 12 hours, twice-a-day controlled release forms of theophylline for 24 hours, once-a-day controlled-release forms of theophylline for 36 hours
9. Subjects who are able to discontinue the following medications for the specified minimum time intervals prior to the run-in period and for the remainder of the study: oral and parenteral corticosteroids for 1 month and oral short-acting beta agonists for 12 hours
10. Subjects who are able and willing to give their written informed consent to participate in the study.

    **********************************************************

    Exclusion Criteria:
11. Female Subjects who are pregnant or breastfeeding
12. Subjects who have life-threatening asthma in the last 10 years, as defined as a history of asthma episode(s) requiring intubation, and/or associated with hypercapnoea; respiratory arrest or hypoxic seizures, asthma-related syncopal episodes(s), or hospitalizations within the past year or during the run-in period
13. Subjects with evidence or history of clinically significant disease or abnormality including congestive heart failure, uncontrolled hypertension, uncontrolled coronary artery disease, myocardial infarction, or cardiac dysrhythmia. In addition, historical or current evidence of significant hematologic, hepatic, neurologic, psychiatric, renal, or other diseases that in the opinion of the investigator, would put the patient at risk through study participation, or would affect the study analyses if the disease exacerbated during the study
14. Subjects with a hypersensitivity to any sympathomimetic drug (e.g. Salmeterol or salbutamol/albuterol) or any inhaled, intranasal or systemic corticosteroid therapy
15. Subjects who are on other medications with the potential to affect the course of asthma or to interact with sympathomimetic amines (e.g. beta blockers, oral decongestants, benzodiazepines, digitalis, phenothiazines, polycyclic antidepressants, monoamine oxidase inhibitors)
16. Subjects with a viral or bacterial upper or lower respiratory tract infection or sinus or middle ear infection within 4 weeks prior to the screening visit or during the run-in period
17. Subjects with any factors (e.g. infirmity, disability, or geographic location) that the investigator feel would likely limit the patient's compliance with the study protocol or scheduled clinic visits
18. Subjects who have used any investigational drug in any clinical trial within 1 month of receiving the first dose of OT329 Solis™ study medication
19. Subjects who cannot communicate reliably or who are unlikely to co-operate with the requirements of the study, in the opinion of the Investigator
20. Subjects with a milk protein allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 879 (Actual)
Dates: Start 2014-09; Primary Completion 2015-05 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rick Fuller, MD FRCP, Study Director — Oriel Therapeutics
Locations (44):
- United States (44):
  - Oriel Investigative Site, Goodyear, Arizona
  - Oriel Investigative Site, Tempe, Arizona
  - Oriel Investigative Site, Anaheim, California
  - Oriel Investigative Site, Los Angeles, California
  - Oriel Invetigative Site, Los Angeles, California
  - Oriel Investigative Site, Mission Viejo, California
  - Oriel Investigative Site, Centennial, Colorado
  - Oriel Investigative Site, Clearwater, Florida
  - Oriel Investigative Site, Coral Gables, Florida
  - Oriel Investigative Site, Homestead, Florida
  - Oriel Investigative Site, Jupiter, Florida
  - Oriel Investigative Site, Kissimee, Florida
  - Oriel Investigative Site, Miami, Florida
  - Oriel Investigative Site, New Port Richie, Florida
  - Oriel Investigative Site, Orlando, Florida
  - Oriel Investigative Site, Tallahassee, Florida
  - Oriel Investigative Site, Lawrenceville, Georgia
  - Oriel Investigative Site, Iowa City, Iowa
  - Oriel Investigative Site, North Dartmouth, Massachusetts
  - Oriel Therapeutics Site, Minneapolis, Minnesota
  - Oriel Investigative Site, St Louis, Missouri
  - Oriel Investigative Site, Bellevue, Nebraska
  - Oriel Investigative Site, Omaha, Nebraska
  - Oriel Investigative Site, Skillman, New Jersey
  - Oriel Investigative Site, Albuquerque, New Mexico
  - Oriel Investigative Site, New York, New York
  - Oriel Investigative Site, Charlotte, North Carolina
  - Oriel Investigative Site, Raleigh, North Carolina
  - Oriel Investigative Site, Winston-Salem, North Carolina
  - Oriel Investigative Site, Cincinnati, Ohio
  - Oriel Investigative Site, Middleburg Heights, Ohio
  - Oriel Investigative Site, Toledo, Ohio
  - Oriel Investigative Site, Oklahoma City, Oklahoma
  - Oriel Investigative Site, Eugene, Oregon
  - Oriel Investigative Site, Medford, Oregon
  - Oriel Investigative Site, Portland, Oregon
  - Oriel Investigative Site, Providence, Rhode Island
  - Oriel Investigative Site, Warwick, Rhode Island
  - Oriel Investigative Site, Rock Hill, South Carolina
  - Oriel Investigative Site, Austin, Texas
  - Oriel Investigative Site, Houston, Texas
  - Oriel Investigative Site, Plano, Texas
  - Oriel Investigative Site, Richmond, Virginia
  - Oriel Investigative Site, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: Yes
Results delayed pending FDA review/approval of drug.

REFERENCES:
- [Derived] Longphre MV, Getz EB, Fuller R. Clinical Bioequivalence of OT329 SOLIS and ADVAIR DISKUS in Adults with Asthma. Ann Am Thorac Soc. 2017 Feb;14(2):182-189. doi: 10.1513/AnnalsATS.201606-436OC. PMID 27849125

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1526 Patients with asthma were screened at 48 clinical sites
Pre-assignment Details: 647 Failed screening (42%)
  * 239 failed because they did not have 40-85% pred FEV1
  * 240 failed because they were not >15% reversible with albuterol
  * 168 failed for other inclusion/exclusion criteria
Period: Overall Study
Arm/Group | OT329 Solis | Advair Diskus | Placebo
Started | 418 | 419 | 42
Completed Day 1 | 418 | 419 | 42
Completed | 395 | 406 | 37
Not Completed | 23 | 13 | 5
Not completed — Adverse Event | 6 | 1 | 2
Not completed — Death | 0 | 1 | 0
Not completed — Lost to Follow-up | 12 | 9 | 0
Not completed — Physician Decision | 2 | 0 | 1
Not completed — Withdrawal by Subject | 3 | 2 | 2

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT)
Groups:
- Total: Total of all reporting groups
Arm/Group | OT329 Solis | Advair Diskus | Placebo | Total
Number analyzed (Participants) | 418 | 419 | 42 | 879
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.9 (14.52) | 43.3 (14.26) | 43.2 (15.25) | 43.6 (14.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 274 | 251 | 30 | 555
  Male | 144 | 168 | 12 | 324
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 122 | 118 | 9 | 249
  Not Hispanic or Latino | 296 | 301 | 33 | 630
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 0 | 4
  Asian | 3 | 4 | 1 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 3 | 0 | 3
  Black or African American | 74 | 89 | 10 | 173
  White | 332 | 308 | 29 | 669
  More than one race | 7 | 13 | 2 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 418 | 419 | 42 | 879
Weight (kg) [Mean (Standard Deviation); unit: Kg] | 88.5 (22.9) | 85.9 (23.1) | 81.0 (17.2) | 86.9 (22.8)
Height (cm) [Mean (Standard Deviation); unit: cm] | 167.5 (9.9) | 169.2 (10.7) | 166.3 (8.3) | 168.2 (10.2)
Body Mass Index [Mean (Standard Deviation); unit: Kg/m^2] | 31.49 (7.61) | 29.91 (7.20) | 29.32 (6.30) | 30.63 (7.40)
Airways Reversibility with Albuterol [Mean (Standard Deviation); unit: % change from pre-albuterol lung functio] — Patients were screened for their airways reversibility following albuterol. Baseline FEV1 was measured then the patient received 360 mcg of albuterol (pMDI), a short-acting adrenergic agonist. Within 30 min of albuterol administration, lung function was measured again. Inclusion Criteria #5 required at least 15% reversibility or improvement in FEV1.
  % change from pre-albuterol lung functio | 30.5 (19.3) | 29.7 (17.5) | 25.9 (13.3) | 29.9 (18.3)

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Serial FEV1-time Curve (AUC 0-12h)
Description: Bioequivalence comparison of lung function (FEV1) for 12 hours after the first dose on Day 1 following OT329 Solis and Advair Diskus treatment. Serial lung function measurements were made pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 10, and 12 hours postdose.
Time Frame: 0-12 hours after dosing on Day 1
Population: Intent-to-treat (ITT)
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | OT329 Solis | Advair Diskus | Placebo
Number analyzed (Participants) | 418 | 419 | 42
Liters | 29.610 (9.044) | 30.151 (9.107) | 27.270 (7.710)
Statistical Analysis 1: Comparison: OT329 Solis vs Advair Diskus; Primary analyses were conducted on BL subtracted values (pre-dose - post-dose). The two one-sided tests method of interval analysis is standard for bioequivalence testing and employs 2 sets of one-sided hypotheses as follows, performed at the 5% alpha level: H01: uT-uR < -0.20 uR vs. Ha1: -0.20 uR </= uT- uR (the lower tail) and H02: uT-uR >0.25 uR vs. Ha2: uT- uR </=0.25 uR (the upper tail) When uT is the LSM SOLIS, uR is the LSM of ADVAIR DISKUS; Test type: Equivalence — Equivalence test compares the Test/Reference with confidence bounds set at standard 80-125%. Superiority test compares Test with Placebo (p<0.05) Superiority test compares Reference with Placebo (p<0.05) (p<0.05); p < 0.05, ANCOVA; Test/Reference = 1.0799, 90% CI 2-sided [.8 to 1.25]; Day 1 superiority to placebo: Solis vs. Placebo p=0.004 Advair vs. Placebo p=0.012

2. Primary Outcome: FEV1 Trough
Description: Bioequivalence comparison of trough lung function (FEV1) after 4 weeks of treatment with OT329 SOLIS or ADVAIR DISKUS.
Time Frame: Post-4 weeks of treatment
Population: Intent-to-Treat
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | OT329 Solis | Advair Diskus | Placebo
Number analyzed (Participants) | 395 | 406 | 37
Liters | 2.516 (0.792) | 2.579 (0.774) | 2.323 (0.736)
Statistical Analysis 1: Comparison: OT329 Solis vs Advair Diskus; Same as the Day 1 analyses; Test type: Equivalence — Standard bioequivalence 90% confidence bounds set at 0.8-1.25; p < 0.05, ANOVA; Test/Reference = 1.0475, 90% CI 2-sided [.8 to 1.25]; Week 4 superiority to placebo: Solis vs. Placebo p=0.019 Advair vs. Placebo p=0.035

3. Secondary Outcome: Number of Participants With Adverse Events
Time Frame: From Screen (Day -28) until 1 week post last treatment
Population: One subject who was assigned OT329 SOLIS received placebo treatment kit in error. The mistake was discovered on Day 1 and the patient was removed from the study. The patient was included in the OT329 SOLIS group for the intent-to-treat analysis but was put in the Placebo group for the Safety analysis as defined by the Statisical Analysis Plan.
Measure: Count of Participants; unit: Participants
Arm/Group | OT329 Solis | Advair Diskus | Placebo
Number analyzed (Participants) | 417 | 418 | 43
Participants | 67 | 66 | 7

ADVERSE EVENTS:
Time Frame: Adverse events were collected from time of consent until 1 week post last treatment, up to 5 weeks. Adverse events from screen failed subjects are omitted.
Description: Treatment emergent adverse events are reported from Day 1 of treatment.
Arm/Group | OT329 Solis | Advair Diskus | Placebo
All-Cause Mortality (participants affected / at risk) | 0/417 | 1/419 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/417 | 2/419 | 0/43
Other Adverse Events (participants affected / at risk) | 52/417 | 47/419 | 7/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OT329 Solis (N=417) | Advair Diskus (N=419) | Placebo (N=43)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) — Fatal heart attack
H. pylori infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — H. pylori gastrointestinal infection leading to hospitalization
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OT329 Solis (N=417) | Advair Diskus (N=419) | Placebo (N=43)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 8 (8) | 6 (6) | 1 (1)
Sinusitis (Infections and infestations) | 4 (4) | 4 (4) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 7 (7) | 5 (5) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 4 (4) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 8 (8) | 13 (13) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 6 (6) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
One patient was randomized to OT329 SOLIS treatment but was given a Placebo kit in error. They are included in the SOLIS group for the efficacy analysis and in the Placebo group for the safety analysis as dictated by the Statistical Analysis Plan.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No